CLINICAL TRIAL: NCT00552435
Title: Phase 2 Study of Micropulse 810nm Diode Laser Photocoagulation for Treatment of Diffuse Diabetic Macular Edema
Brief Title: Micropulse 810 Nanomolar (nm), Diode Laser for Diffuse Diabetic Macular Edema
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Federal University of Sao Paulo, Vision Institute Department of Ophthalmology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MP-001
Record Dates: First submitted 2007-10-31; First posted 2007-11-02 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-05

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental): Micropulse 810nm diode laser
  Interventions: Device: Laser photocoagulation
- 2 (Active Comparator): Argon laser photocoagulation
  Interventions: Device: Laser photocoagulation

INTERVENTIONS:
Device: Laser photocoagulation — Laser therapy is applied using a slit lamp and specific laser contact lens.

SUMMARY:
Objective: To compare micropulse 810nm diode laser photocoagulation versus argon laser photocoagulation for treatment of diabetic macular edema. Micropulse laser technique will be determined by an initial clinical trial comparing single versus double density laser photocoagulation techniques for treatment of diabetic macular edema.The single density is based on the Early Treatment Diabetic Retinopathy Study (ETDRS) grid photocoagulation technique and the double density increases the number of spots.

Methods: Patients with diabetic macular edema will be assigned to receive either micropulse 810nm diode laser photocoagulation or argon laser photocoagulation therapy. First, in a smaller clinical trial, patients will be assigned to single or double density micropulse 810nm diode laser to determine best strategy for this therapy. Visual acuity, fundus photographs and fluorescein angiography, and optical coherence tomography measurements , autofluorescence and mfERG were obtained at baseline and at 1, 3 and 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus (type 1 or 2)
* Diabetic macular edema in study eye associated to diabetic retinopathy
* Diffuse macular edema defined as macular thickening determined by biomicroscopy and fluorescein angiography.
* Best corrected visual acuity between 34 (20/200) and 68 letters (20/50).
* Macular thickness greater than 300 mcm on OCT.

Exclusion Criteria:

* Uncontrolled systemic disease
* Start of medical therapy for diabetes or change in treatment from oral to insulin four months before initial visit.
* HbA1c levels greater than 10%
* Presence of retinal venous occlusion, cystoid macular edema,or other condition that would contribute to macular edema.
* Presence of epiretinal membrane
* Presence of vitreomacular traction in the study eye.
* Neovascularization of disc or elsewhere in the study eye.
* History or presence of choroidal neovascularization in the study eye.
* Presence of rubeosis irides in the study eye.
* Eye opacity that interfere with clinical documentation and photography.
* Intra-ocular surgery 90 days before initial visit.
* Scheduled surgery for study eye.
* Patients with known allergies to fluorescein.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-03; Primary Completion 2008-11 (Estimated); Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
Macular thickness measured by optical coherence tomography (OCT) | 12 months

SECONDARY OUTCOMES:
Safety profile | 12 months
Selectivity of laser therapy (autofluorescence and mfERG) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Cardillo, Principal Investigator — Federal University of Sao Paulo- Department of Ophthalmology
Locations (1):
- Vision Institute, Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Lavinsky D, Cardillo JA, Melo LA Jr, Dare A, Farah ME, Belfort R Jr. Randomized clinical trial evaluating mETDRS versus normal or high-density micropulse photocoagulation for diabetic macular edema. Invest Ophthalmol Vis Sci. 2011 Jun 17;52(7):4314-23. doi: 10.1167/iovs.10-6828. PMID 21345996